CLINICAL TRIAL: NCT04127734
Title: Treatment of AnastomotiC Leakage After Rectal Cancer Resection. TENTACLE Rectum Study
Brief Title: Treatment of Anastomotic Leakage After Rectal Cancer Resection
Acronym: TENTACLE:R
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-5849
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Anastomotic Leak Rectum; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: The efficacy of various interventions for anastomotic leakage after rectal cancer resection are investigated — Investigated interventions comprise conservative, radiological, endoscopic and surgical (including stoma formation) interventions

SUMMARY:
The TENTACLE: Rectum study is a multinational retrospective cohort study that includes patients with anastomotic leakage after rectal cancer resection.

The study aims to develop an anastomotic leakage severity score and to evaluate the efficacy of different treatments of anastomotic leakage.

DETAILED DESCRIPTION:
Rationale:

Anastomotic leakage occurs in up to 20% after low anterior resection for rectal cancer. It is a severe complication with high associated morbidity, ICU admission, prolonged hospital stay and need for reinterventions and readmissions. Anastomotic leakage is independently associated with the risk of local recurrence and reduced long term survival. Most literature focusses on incidence and predictive factors. Remarkably, there is almost no data on the efficiency of different treatments of anastomotic leakage after low anterior resection.

Anastomotic leakage after rectal cancer resection is generally underreported, mainly due to subclinical leaks below a diverting stoma. However, up to 50% of the leaks do not heal with fecal diversion alone, especially not in an irradiated field, related to a competent sphincter which hampers adequate drainage of the presacral abscess. Late diagnosis of 'reactivated' leaks after stoma reversal is not an infrequent phenomenon. Chronic sinus, gluteal abscess, and fistula formation have been reported in up to 10%, and permanent stoma rates around 20%, both having significant impact on quality of life.

Examples of factors that may influence the severity and chance of healing of the anastomotic leakage are: timing of diagnosis, degree of systemic inflammatory response, etiology (e.g. ischemia of the afferent loop), degree of dehiscence and retraction, location of the leak (e.g. circular staple line, blind loop), whether or not a diverting stoma is in place, and extent of abdominal contamination. However, little is known about to what extent these and other factors contribute to anastomotic leakage severity and chance of healing. In addition, it is not known which anastomoses are likely to be preserved by which type of treatment, and which anastomotic failures require redo surgery at a certain time frame.

Primary study objectives

1. To investigate which factors contribute to anastomotic leakage severity and to compose an evidence based anastomotic leakage severity score, in which clinically relevant subgroups will be explored (e.g. diversion or not), as well as different clinical settings (e.g. leak diagnosis within or beyond 90 days postoperatively).
2. To evaluate the effects of different treatment approaches on all different pre-specified outcome parameters, stratified for severity score, anatomical characteristics of leakages and timing of diagnosis of leakage.

Study design:

International multicenter retrospective cohort study.

Study population:

Adult patients with anastomotic leakage after low anterior resection for rectal cancer.

Primary outcome parameter:

1-year stoma-free survival.

Secondary outcome parameters:

ICU length of stay, mortality, comprehensive complications index, total number of reinterventions (surgical, radiological, endoscopic) within one year, total number of unplanned readmissions within one year, total hospital stay during one year, total time of having a stoma until one year, stoma present at one year, type of stoma present at one year (diverting, permanent), secondary leakage related complications (extrapelvic abscess, cutaneous fistula, vaginal fistula, bladder fistula, small bowel, ureteric fibrosis with hydronephrosis), hospital related costs.

Sample size calculation:

Inclusion of 980 patients will be sufficient to analyze primary study objective 1 and this is 1246 patients for primary study objective 2. Therefore, the aim is to include at least 1246 patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Cancer located in the rectum, defined according to the international definition of the rectum consensus [D'Souza 2019];
* Rectal cancer resection with primary anastomosis (with or without diverting loop ileostomy) for either primary cancer, completion after local excision or salvage resection for regrowth after watch & wait or local excision;
* Postoperative anastomotic leakage according to the following definition: "a breach in a surgical join between two hollow viscera, with or without active leak of luminal contents" [Peel 1991].

Exclusion Criteria:

* Rectal resection for benign disease;
* Rectal resection for recurrent rectal cancer after previous low anterior resection or other primary malignancies;
* Multivisceral resection (lateral lymph node dissection can be included)
* Emergency resection;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult rectal cancer patients who have been operated between January 2014-December 2018 will be retrospectively analyzed and evaluated for an anastomotic leakage. All patients with an anastomotic leakage diagnosed within one year from primary surgery are suitable for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1246 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
1-year stomafree survival | 1 year
  Survival of the patient and absence of a stoma

SECONDARY OUTCOMES:
ICU length of stay | 1 year
  Length of stay in the intensive care unit
1 year mortality | 1 year

OTHER OUTCOMES:
Comprehensive complications index | 1 year
  According to Clavien
Readmission rate | 1 year
  Readmission to the hospital after discharge
Reintervention rate | 1 year
  Total number of reinterventions (radiological, surgical, endoscopic)
Hospital length of stay | 1 year
  Total days in the hospital
Stoma time | 1 year
  Total time of having a stoma
Type of stoma present at 1 year | 1 year
Secondary leak related complication rate | 1 year
  extrapelvic abscess, cutaneous fistula, vaginal fistula, bladder fistula, small bowel fistula, ureteric fibrosis with hydronefrosis
Hospital related costs | 1 year
  Costs of hospital/ICU stay and interventions/diagnostics

CONTACTS AND LOCATIONS:
Overall Officials: Hans de Wilt, MD, PhD, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
Planning to share IPD with collaborators if interesting research questions are submitted to the study steering committee.
  Specifics will be determined in study meetings in the nearby future.